CLINICAL TRIAL: NCT00210821
Title: A Comparison of Topiramate Versus Amitriptyline in Migraine Prophylaxis
Brief Title: Comparing the Safety and Effectiveness of Topiramate With the Safety and Effectiveness of Amitriptyline in Preventing Migraine Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR004666
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-05

CONDITIONS: Migraine; Headache
Keywords: migraine; headache; analgesics; prophylaxis; prevention
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of two treatment regimens in preventing migraines. The antidepressant amitriptyline has been used successfully to prevent migraine headaches.

DETAILED DESCRIPTION:
People who suffer from migraines have many prescription medications to choose from, both to treat the migraine and to prevent it from starting. However, many patients have not had success in finding the drug that helps them best. Amitriptyline, an antidepressant, has been used successfully for many years to prevent migraine headaches. This study will compare the effectiveness of amitriptyline with the effectiveness of topiramate, an anti-seizure drug, in preventing migraines. The safety of both drugs will also be assessed. The objective of the study is to demonstrate that topiramate will be at least as effective as amitriptyline in preventing migraines. During the first 4 weeks of the study, topiramate or amitriptyline will be increased by 25 mg per week up to a total dose of 100 mg per day or up to the maximum tolerated dose, whichever is less. Treatment will continue at 100 mg per day for 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Migraine headache for at least 6 months, with 3 to 12 headaches a month for the previous 3 months
* no more than 15 headache days in the previous month before study start
* no heart rhythm problems or neurologic problems
* women must not be pregnant and must use birth control

Exclusion Criteria:

* Cannot have failed at least 2 previous trials of migraine prevention drugs
* cannot have failed a previous trial of topiramate or amitriptyline
* no cluster headaches
* no migraine with aura without headache
* no pain that is worse than the migraine pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2004-02; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average monthly migraine episode rate.

SECONDARY OUTCOMES:
Change in average monthly rate of days with migraine headache; change in average monthly rate of headache (migraine & non-migraine) days; change in average monthly rate of acute abortive medications; weight changes; quality of life assessments

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Comparison of Topiramate Versus Amitriptyline in Migraine Prophylaxis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=617&filename=CR004666_CSR.pdf